CLINICAL TRIAL: NCT00738816
Title: The Effect of Systematic Medication Review in Elderly Patients Admitted to an Orthopedic Department.
Brief Title: Effect of Systematic Medication Review in Elderly Patients Admitted to an Orthopedic Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Marianne Lisby, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Klinfarm
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Elderly
Keywords: Medication review; Patient; Safety; Drug; Prescriptions; Drug-use

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other): Systematic medication review
  Interventions: Other: Systematic medication review and advisory notes

INTERVENTIONS:
Other: Systematic medication review and advisory notes — Within 24 hours of admission a pharmacist retrieve medication histories from patients included in the intervention group. Medication histories will be obtained from - medical records, medication charts, patients electronical medication profile, interview with patients and if necessary contact to the patients general practitioner. The obtained medication history will be discussed with a physician specialized in pharmacology and an advisory note with suggested changes to the patients medication is added to the medical record. The orthopedic physicians are not obliged to follow the suggested changes

SUMMARY:
Elderly patients have a higher risk of experiencing adverse drug events due to an age related increase in morbidity and medication use. Inappropriate or wrong medication use among elderly patients acutely admitted to hospitals is assumed to result in earlier contact to general practitioner, emergency departments and re-admissions if not corrected during hospital admission. It is therefore our hypothesis that a systematic medication review conducted by pharmacists and physicians specialized in pharmacology will increase time to first unscheduled physician contact (general practitioner, emergency departments, ambulatory care and re-admissions) after discharge from hospital from an average of 21days to 25 days. Further, the following secondary outcome parameters will be measured at discharge and within 3-month follow-up:

* length of in-hospital stay
* number of contacts to general practitioner 30 days after discharge, that resulted in medication changes
* number of re-admissions at 3-month
* number of death at 3-month
* number of contact to primary health care at 3-month
* patients self-experienced quality of health(EQ-5D) 3-month

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* expected admission time of more than 24 hours
* acute admission

Exclusion Criteria:

* Psychotic patients
* Moribund patients
* Suicidal patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Time to first unscheduled physician contact(general practitioner,emergency department, ambulatory care or re-admission to hospital) after discharge from the Orthopaedic Department | January 2010

SECONDARY OUTCOMES:
Admission time | October 2009

CONTACTS AND LOCATIONS:
Overall Officials: Nielsen Lars Peter, Assoc. Prof., Principal Investigator — Aarhus University Hospital, Denmark
Locations (1):
- Regional hospital, Randers, Randers, Central Jutland, Denmark

REFERENCES:
- [Background] Holland R, Desborough J, Goodyer L, Hall S, Wright D, Loke YK. Does pharmacist-led medication review help to reduce hospital admissions and deaths in older people? A systematic review and meta-analysis. Br J Clin Pharmacol. 2008 Mar;65(3):303-16. doi: 10.1111/j.1365-2125.2007.03071.x. Epub 2007 Dec 17. PMID 18093253
- [Background] Lau HS, Florax C, Porsius AJ, De Boer A. The completeness of medication histories in hospital medical records of patients admitted to general internal medicine wards. Br J Clin Pharmacol. 2000 Jun;49(6):597-603. doi: 10.1046/j.1365-2125.2000.00204.x. PMID 10848724
- [Background] Glintborg B, Andersen SE, Dalhoff K. Drug-drug interactions among recently hospitalised patients--frequent but mostly clinically insignificant. Eur J Clin Pharmacol. 2005 Oct;61(9):675-81. doi: 10.1007/s00228-005-0978-6. Epub 2005 Oct 19. PMID 16047138
- [Background] Page RL 2nd, Ruscin JM. The risk of adverse drug events and hospital-related morbidity and mortality among older adults with potentially inappropriate medication use. Am J Geriatr Pharmacother. 2006 Dec;4(4):297-305. doi: 10.1016/j.amjopharm.2006.12.008. PMID 17296535
- [Background] Vira T, Colquhoun M, Etchells E. Reconcilable differences: correcting medication errors at hospital admission and discharge. Qual Saf Health Care. 2006 Apr;15(2):122-6. doi: 10.1136/qshc.2005.015347. PMID 16585113